CLINICAL TRIAL: NCT05531669
Title: Effect of PLAY Project Intervention Program on Children With Autism Spectrum Disorder: A Multi-center, Randomized Control Study in China
Brief Title: Effect of PLAY Project Intervention Program on Children With ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Fuzhou Children's Hospital of Fujian Medical University (Unknown); Third Affiliated Hospital of Zhengzhou University (Other); Shenzhen Hospital of Southern Medical University (Other); Children's Hospital of Zhejiang University School of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJPLAY
Record Dates: First submitted 2022-08-31; First posted 2022-09-08 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; PLAY Project; functional developmental level
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): the study group will receive 12 months of Play Project + Parental Education intervention
  Interventions: Behavioral: PLAY Project; Behavioral: Parental Education
- control group (Active Comparator): the control group will receive Parental Education intervention in the first 6 months, and then receive Play Project + Parental Education intervention in the next 6 months
  Interventions: Behavioral: PLAY Project; Behavioral: Parental Education

INTERVENTIONS:
Behavioral: PLAY Project — PLAY consultants coached caregivers monthly for 12 months to improve caregiver-child interaction using videotape and written feedback within a developmental framework.
Behavioral: Parental Education — Each study center provides welcome course and parent guide for families with ASD children monthly.

SUMMARY:
The objective of this study is to evaluate the effectiveness of the Play and Language for Autistic Youngsters (PLAY) Project Home Consultation model to improve parent-child interaction, child development, and autism symptomatology in young children with autism spectrum disorders (ASDs) in China.

DETAILED DESCRIPTION:
The present multi-center randomized controlled trial will recruit 200 children with ASD aged 18 months to 6 years from 5 hospitals including Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Fuzhou Children's Hospital of Fujian Medical University, The Third Affiliated Hospital of Zhengzhou University, Shenzhen Hospital of Southern Medical University and Children's Hospital of Zhejiang University School of Medicine from 2022.8 to 2023.1.Children who meet the inclusion criteria will be stratified by ASD severity, age and gender and randomly assigned (1:1) to either study group or control group. Using the waitlist-control group design, the study group will receive 12 months of Play Project + Parental Education intervention, the control group receive Parental Education intervention in the first 6 months, and then receive Play Project + Parental Education intervention in the next 6 months. Pre-, 6th month and post- assessments for both groups will be conducted, including Diagnostic and Statistical Manual of Mental Disorders fifth edition (DSM-Ⅴ), Autism Diagnostic Observation Schedule-Second Edition (ADOS-2), Social Communication Questionnaire (SCQ), Child Autism Rating Scale (CARS), Gesell Developmental Schedules (GDS) for children; Raven's Standard Progressive Matrices (SPM), Hamilton Depression Scale (HAMD) and Parenting Stress Index-Short Form (PSI-SF) for parents, Maternal Behavior Rating Scale (MBRS) and Pivotal Behavior Rating Scale (PBRS).

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 months to 6 years old at the time of enrollment, no gender requirement;
2. Children who were diagnosed with autism spectrum disorder in 5 research centers, meet the diagnostic criteria by Diagnostic and Statistical Manual of Mental Disorders fifth edition (DSM-Ⅴ), and the Autism Diagnostic Observation Schedule-Second Edition (ADOS-2).
3. Complete pre-assessments in outpatient clinics, including: Diagnostic and Statistical Manual of Mental Disorders fifth edition (DSM-Ⅴ), Autism Diagnostic Observation Schedule-Second Edition (ADOS-2), Social Communication Questionnaire (SCQ), Child Autism Rating Scale (CARS), Gesell Developmental Schedules (GDS) for children; Raven's Standard Progressive Matrices (SPM), Hamilton Depression Scale (HAMD) and Parenting Stress Index-Short Form (PSI-SF) for parents.
4. Parents agreed to participate in the study provided written informed consent at recruitment.

Exclusion Criteria:

1. High functioning ASD children with abnormal social communication but high language level. Language development quotient>85 in GDS;
2. Suffering from:

   1. hereditary diseases, such as Rett syndrome, Fragile X syndrome, trisomy 21 or tuberous sclerosis;
   2. abnormal vision or hearing impairment;
   3. movement disorders, such as cerebral palsy;
   4. epilepsy;
3. Receive 7 hours or more per week of 1:1 intensive intervention, such as Applied Behavior Analysis (ABA), Parent-Implemented Language training, etc.
4. Parents scoring <90 by SPM, or report being severely depressed by HAMD, will be excluded from the study.

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Diagnostic and Statistical Manual of Mental Disorders fifth edition (DSM-Ⅴ) in ASD children | baseline, 6th-months, 12th-months
  DSM-5 provides core symptom domain severity levels based on the level of support needed for individual functioning, in addition to specifiers which offer descriptions of common co-occurring non-ASD impairments (i.e., intellectual impairments, language deficits, medical and psychiatric conditions, etc.)
Changes in Autism Diagnostic Observation Schedule-Second Edition (ADOS-2) in ASD children | baseline, 6th-months, 12th-months
  ADOS-2 is a standardized diagnostic instrument designed to assess communication, social interaction, play skills, and restrictive and repetitive behaviors (RRB). The ADOS-2 can be used with individuals at a wide range of developmental and language levels: Module 1 for use with children who do not consistently use phrase speech; Module 2 for children who use phrase speech, but are not verbally fluent; Module 3 for verbally fluent children and young adolescents; and Module 4 for verbally fluent older adolescents and adults. The calibrated severity scores (CSS) have been created for Autism Diagnostic Observation Schedule, 2nd edition (ADOS-2), Modules 1-4 as a metric of the relative severity of autism-specific behaviors.
Changes in Child Autism Rating Scale (CARS) in ASD children | baseline, 6th-months, 12th-months
  CARS assesses the child on a scale from 1 to 4 in each of 15 dimensions or symptoms. A total score of at least 30 strongly suggests the presence of autism. Children with score between 30 and 36 have mild-to-moderate autism while those with score between 37 and 60 have severe autism.
Changes in Social Communication Questionnaire (SCQ) in ASD children | baseline, 6th-months, 12th-months
  The Social Communication Questionnaire (SCQ) is one of the standardized screening tools used to identify ASD. It contains 40 questions about reciprocal social interaction, communication, and repetitive/stereotypic behavior. Each yes/no item (scored as 1 or 0, respectively) indicates the presence or absence of developmentally inappropriate behaviors. Scores range between 0 and 33 for individuals without verbal speech and from 0 to 39 for verbal individuals. In addition, higher scores indicate more worrisome behaviors, and a cutoff score of ≥15 points is established as indicating a risk of ASD.
Changes in Gesell Developmental Schedules (GDS) in ASD children | baseline, 6th-months, 12th-months
  Developmental and language assessment，A subscale DQ less than 76 points indicates a developmental delay, a quotient between 76 and 85 points is slightly below the threshold for developmental delay, and a quotient greater than or equal to 86 points indicates normal development. Performance in each area was recorded as an equivalent developmental age in months. Developmental quotients were calculated by comparing the children's performance equivalent age and their chronological age at the time of administration (DQ=developmental age / chronological age x 100).
Changes in Pivotal Behavior Rating Scale (PBRS) in ASD children | baseline, 6th-months, 12th-months
  The PBRS is a key outcome measure of contingent, reciprocal, social interactions. PBRS measures two components of interactive behavior - Attention and Initiation. The child's primary caregiver is asked to play with the child for 7 ½ minutes using a standard set of toys. Independent raters, blind to subject status, review a videotape of the session and score the child's behavior on seven items: attention to activity; persistence (practice/problem solving); involvement (vs. distractibility); cooperation; initiate activities; joint attention; and affect (emotional state during play).
Changes in Maternal Behavior Rating Scale (MBRS) in the interaction between ASD children and their parents | baseline, 6th-months, 12th-months
  MBRS is a video rating scale that assesses four Interactive Style Factors including: Responsive/Child Oriented; Affect/Animation; Achievement Orientation; and Directiveness (Aim 1, Outcomes 1-3). Factors are assessed by rating twelve (5 point Likert-scaled) items during a 7 ½ minute video of typical parent-child play with toys.

SECONDARY OUTCOMES:
Raven's Standard Progressive Matrices (SPM) | baseline
  SPM is an intelligence quotient(IQ) screen to ensure that parents have the cognitive/verbal skills to properly translate information into action. Parents scoring less than 90 will be excluded from the study.
Hamilton Depression Scale (HAMD) | baseline
  HAMD assesses whether parents have the emotional functionality needed to deliver the intervention. Parents who report being severely depressed will be excluded from the study.
Changes in Parenting Stress Index-Short Form (PSI-SF) in parents of ASD children | baseline, 6th-months, 12th-months
  Parenting stress is assessed using the PSI-SF, consists of 36 items.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Hao, doctor, Principal Investigator — Tongji Hospital
Locations (5):
- China (5):
  - Fuzhou Children's Hospital of Fujian Medical University, Fuzhou, Fujian
  - Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hyman SL, Levy SE, Myers SM; COUNCIL ON CHILDREN WITH DISABILITIES, SECTION ON DEVELOPMENTAL AND BEHAVIORAL PEDIATRICS. Identification, Evaluation, and Management of Children With Autism Spectrum Disorder. Pediatrics. 2020 Jan;145(1):e20193447. doi: 10.1542/peds.2019-3447. Epub 2019 Dec 16. PMID 31843864
- [Background] Gnanavel S, Robert RS. Diagnostic and statistical manual of mental disorders, fifth edition, and the impact of events scale-revised. Chest. 2013 Dec;144(6):1974. doi: 10.1378/chest.13-1691. No abstract available. PMID 24297138
- [Background] Lord C, Charman T, Havdahl A, Carbone P, Anagnostou E, Boyd B, Carr T, de Vries PJ, Dissanayake C, Divan G, Freitag CM, Gotelli MM, Kasari C, Knapp M, Mundy P, Plank A, Scahill L, Servili C, Shattuck P, Simonoff E, Singer AT, Slonims V, Wang PP, Ysrraelit MC, Jellett R, Pickles A, Cusack J, Howlin P, Szatmari P, Holbrook A, Toolan C, McCauley JB. The Lancet Commission on the future of care and clinical research in autism. Lancet. 2022 Jan 15;399(10321):271-334. doi: 10.1016/S0140-6736(21)01541-5. Epub 2021 Dec 6. No abstract available. PMID 34883054
- [Background] Maenner MJ, Shaw KA, Bakian AV, Bilder DA, Durkin MS, Esler A, Furnier SM, Hallas L, Hall-Lande J, Hudson A, Hughes MM, Patrick M, Pierce K, Poynter JN, Salinas A, Shenouda J, Vehorn A, Warren Z, Constantino JN, DiRienzo M, Fitzgerald RT, Grzybowski A, Spivey MH, Pettygrove S, Zahorodny W, Ali A, Andrews JG, Baroud T, Gutierrez J, Hewitt A, Lee LC, Lopez M, Mancilla KC, McArthur D, Schwenk YD, Washington A, Williams S, Cogswell ME. Prevalence and Characteristics of Autism Spectrum Disorder Among Children Aged 8 Years - Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2018. MMWR Surveill Summ. 2021 Dec 3;70(11):1-16. doi: 10.15585/mmwr.ss7011a1. PMID 34855725
- [Background] Zhou H, Xu X, Yan W, Zou X, Wu L, Luo X, Li T, Huang Y, Guan H, Chen X, Mao M, Xia K, Zhang L, Li E, Ge X, Zhang L, Li C, Zhang X, Zhou Y, Ding D, Shih A, Fombonne E, Zheng Y, Han J, Sun Z, Jiang YH, Wang Y; LATENT-NHC Study Team. Prevalence of Autism Spectrum Disorder in China: A Nationwide Multi-center Population-based Study Among Children Aged 6 to 12 Years. Neurosci Bull. 2020 Sep;36(9):961-971. doi: 10.1007/s12264-020-00530-6. Epub 2020 Jun 30. PMID 32607739
- [Background] Magiati I, Tay X W, Howlin P. Early comprehensive behaviorally based interventions for children with autism spectrum disorders: a summary of findings from recent reviews and meta-analyses [J]. Neuropsychiatry, 2012, 2(6): 543-570.
- [Background] Rogge N, Janssen J. The Economic Costs of Autism Spectrum Disorder: A Literature Review. J Autism Dev Disord. 2019 Jul;49(7):2873-2900. doi: 10.1007/s10803-019-04014-z. PMID 30976961
- [Background] Kodak T, Bergmann S. Autism Spectrum Disorder: Characteristics, Associated Behaviors, and Early Intervention. Pediatr Clin North Am. 2020 Jun;67(3):525-535. doi: 10.1016/j.pcl.2020.02.007. Epub 2020 May 4. PMID 32443991
- [Background] Sanchack KE, Thomas CA. Autism Spectrum Disorder: Primary Care Principles. Am Fam Physician. 2016 Dec 15;94(12):972-979. PMID 28075089
- [Background] Solomon R, Van Egeren LA, Mahoney G, Quon Huber MS, Zimmerman P. PLAY Project Home Consultation intervention program for young children with autism spectrum disorders: a randomized controlled trial. J Dev Behav Pediatr. 2014 Oct;35(8):475-85. doi: 10.1097/DBP.0000000000000096. PMID 25264862
- [Background] Oono IP, Honey EJ, McConachie H. Parent-mediated early intervention for young children with autism spectrum disorders (ASD). Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD009774. doi: 10.1002/14651858.CD009774.pub2. PMID 23633377
- [Background] Hume K, Steinbrenner JR, Odom SL, Morin KL, Nowell SW, Tomaszewski B, Szendrey S, McIntyre NS, Yucesoy-Ozkan S, Savage MN. Evidence-Based Practices for Children, Youth, and Young Adults with Autism: Third Generation Review. J Autism Dev Disord. 2021 Nov;51(11):4013-4032. doi: 10.1007/s10803-020-04844-2. Epub 2021 Jan 15. PMID 33449225